CLINICAL TRIAL: NCT00710125
Title: Phase 1 Study and Dose Seeking Study of an Intravenous Formulation of the Anthracycline Analog GPX-150 in Patients With Solid Tumors
Brief Title: Safety Study of GPX-150 in Patients With Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Gem Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GPX-150-001
Record Dates: First submitted 2008-07-02; First posted 2008-07-04 (Estimated); Last update posted 2014-08-05 (Estimated); Status verified 2014-08

CONDITIONS: Advanced Solid Tumors - Phase 1 Population
MeSH Terms: interventions — 5-imino-13-deoxydoxorubicin; Injections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- GPX-150 for Injection (Experimental): GPX-150 is administered IV on Day 1, followed by a 20 day rest period, every 3 weeks.
  Interventions: Drug: GPX-150 for Injection

INTERVENTIONS:
Drug: GPX-150 for Injection — Escalating doses starting at the dose of 14 mg/m2 and increasing to the dose of 265 mg/m2 will be administered IV once every 3 weeks for up to 8 cycles of treatment. Patients who have previously received an anthracycline are limited to 4 cycles of treatment.
  Other Names: GPX-150; 5-imino-13-deoxy-doxorubicin HCl

SUMMARY:
This is a Phase 1 safety and dose escalation study to define the maximum tolerated dose (MTD) and identify the dose limiting toxicities (DLT) following IV administration of GPX-150 once every 3 weeks. Escalating doses starting at the dose of 14 mg/m2 and increasing to the dose of 265 mg/m2 will be administered IV once every 3 weeks for up to 8 cycles of treatment. Patients who have previously received an anthracycline are limited to 4 cycles of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patient is at least 18 years of age.
* Patient has a histologically or cytologically confirmed diagnosis of solid tumor.
* Patient has progressive disease
* Patient is considered to have incurable disease and is not a candidate for known effective systemic treatment.
* Patient has a performance status of at least 70% on Karnofsky scale.
* Patient has not received any cytotoxic chemotherapy or other investigational agents within 4 weeks of the first treatment in this study (6 weeks for mitomycin or nitrosourea). Patients should receive supportive care as indicated. Patients currently receiving blood transfusions or erythropoiesis-stimulating agents should continue receiving them as per the ASCO guidelines. Patients requiring palliative radiation therapy should complete their course of radiation treatment 4 weeks before the first study treatment.
* Patient may have received unlimited prior hormonal therapy, but this must have been completed at least 4 weeks prior to the first study treatment, and progressive disease documented following withdrawal of hormone therapy. Patient with hormone-refractory prostate cancer on long acting LHRH agents may continue on these agents.
* Patient may have received unlimited prior biological or immunological therapy without limitation, but this must have been completed at least 4 weeks prior to the first study treatment.
* Patient has fully recovered from any previous surgery (at least 4 weeks since major surgery) and radiation therapy (at least 4 weeks since the end of treatment).
* Patient has recovered from reversible toxicity of prior therapy. Permanent and stable side effects or changes are acceptable if ≤ to Grade 2.
* Patient has adequate hematological function as defined by an ANC ≥ 1500, platelets ≥ 100,000/µL, and hemoglobin ≥9.0 gm/dL.
* Patient has adequate organ function defined as a bilirubin ≤ 1.5 times ULN, AST and ALT < 2.5 times the upper limit of normal (ULN, 5.0 times the ULN with liver involvement), serum creatinine <2.0 dL or estimated creatinine clearance ≥ 50 ml/min.
* Patient has an ejection fraction of 110% of the lower limit of institutional normal as determined by resting MUGA scan.
* Patient has an O2 Sat by pulse oximetry of at least 90%.
* Patient has a negative pregnancy test prior to study entry if premenopausal or if less than 12 months after menopause. Premenopausal patients must use a medically effective form of contraception during the treatment period.
* Patient is willing and able to comply with all study protocol requirements. The patient or a legally authorized representative must fully understand all elements of the informed consent and have signed the informed consent according to institutional and federal regulatory requirements.

Exclusion Criteria:

* Patient is pregnant or breast-feeding.
* Patient has a history of hypersensitivity to anthracyclines.
* Patient has received a cumulative dose of doxorubicin that exceeds 300 mg/m2 or a cumulative dose of epirubicin that exceeds 540 mg/m2.
* Patient has received an anthracycline within 6 months prior to entry into the study.
* Patient has brain metastases unless asymptomatic and stable off glucocorticoids.
* Prior history of CHF, myocardial infarction within 6 months prior to enrollment, active ischemic heart disease, or uncontrolled hypertension.
* Patient requires active medical therapy for CHF or arrhythmia.
* Patients with > Grade l motor neuropathy or > Grade 2 sensory neuropathy.
* Patient has participated in a study of any investigational drug within 4 weeks prior to the first study treatment.
* Patient has received chemotherapy, hormonal therapy (with the exception of LHRH for prostate cancer), immunotherapy, biological therapy, or radiotherapy within 4 weeks prior to the first study treatment.
* Patient has had major surgery within 4 weeks of the first study treatment.
* Patient has received G-CSF or GM-CSF within 4 weeks prior to first dose of study drug.
* Patient has baseline laboratory values that are outside normal ranges or those listed (see Inclusion Criteria), which are clinically significant as determined by the investigator.
* Patient has a serious, concurrent medical condition that would limit the patient's ability to complete or comply with the study requirements.
* Patient is unable or unwilling to comply with the contraceptive requirements during the study period.
* Patient has lymphoma.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2008-01; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Define maximum tolerated dose and identify dose limiting toxicities following IV administration of GPX-150 for Injection once every 3 weeks | Every 3 weeks

SECONDARY OUTCOMES:
Pharmacokinetics and any antitumor activity | Every 3 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Raymond J Hohl, MD, PhD, Principal Investigator — University of Iowa
Locations (1):
- University of Iowa Hospital and Clinics, Iowa City, Iowa, United States